CLINICAL TRIAL: NCT03149406
Title: Study of microRNAs in the Evolution of Carotid Plaque. Physiopathological and Therapeutic Interest
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2012_843_0019
Record Dates: First submitted 2017-05-04; First posted 2017-05-11 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: miRNAs; Carotid Plaque

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic patients: in the department with carotid plaque Comparing the expression of miRNAs
  Interventions: Other: Comparing the expression of miRNAs
- Asymptomatic patients: in consultation with carotid plaque Comparing the expression of miRNAs
  Interventions: Other: Comparing the expression of miRNAs

INTERVENTIONS:
Other: Comparing the expression of miRNAs — by PCR, in symptomatic and asymptomatic carotid plaques.

SUMMARY:
Carotid stenosis of atherosclerotic origin may be responsible for stroke, which is one of the most important causes of morbidity and mortality in the Western world

DETAILED DESCRIPTION:
Carotid stenosis of atherosclerotic origin may be responsible for stroke, which is one of the most important causes of morbidity and mortality in the Western world. The constitution of the atheroma plaque is linked to the deregulation of several biological phenomena, including angiogenesis, adipogenesis, inflammatory response, lipid metabolism and oxidative stress. In addition to its anatomical and physiological characteristics, the notion of plate stability is of paramount importance for clinical implications. This stability depends largely on the biological composition of the plate. A vulnerable or unstable plaque often has a large lipid body consisting of foam cells (macrophages laden with oxidized LDL) with a thin fibrous screed consisting of smooth muscle cells (CML), collagen fibers and extracellular matrix. This plaque is also made up of numerous inflammatory cells including macrophages, rich vascularization and intraplate hemorrhage. Although the cell composition of the unstable plate is still relatively established, its molecular analysis remains little known.

The benefit of carotid surgery in asymptomatic patients with stenosis greater than 70% is increasingly controversial given the moderate risk of spontaneous stroke under optimal medical treatment. This annual average risk is less than 5%. Thus, the discovery of an original and innovative biomarker, predictive of plate rupture, would define the patients most at risk, who benefit most from this surgery.

ELIGIBILITY:
Inclusion Criteria:

* Any adult with a carotid thrombo endarterectomy,
* affiliated to a social security scheme,
* informed of the study and not opposed to it.

Exclusion Criteria:

* Any person benefiting from an iterative carotid surgery,
* or refusing to participate in the study,
* or not being able to express its consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic patients in the service, and asymptomatic in consultation with carotid atheroma plaque
Sampling Method: Non-Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2012-12-26 (Actual); Primary Completion 2020-12-26 (Estimated); Study Completion 2020-12-26 (Estimated)

PRIMARY OUTCOMES:
Analysis of the miRNAs | 3 years
  by PCR of the composition of the atheroma plaque

CONTACTS AND LOCATIONS:
Overall Officials: Thierry REIX, PhD, Principal Investigator — CHU AMIENS-PICARDIE
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France